CLINICAL TRIAL: NCT04601194
Title: Study Title: Goal Elicitation, Treatment Prioritization, & Electronically-Practiced Discussion - Pilot Study
Brief Title: Goal Elicitation, Treatment Prioritization, & Electronically-Practiced Discussion for Psychiatry
Acronym: GET-PrEPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Florida (Other); Eskenazi Health (Other)
Responsible Party: Principal Investigator, Michelle Salyers, Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010326129; 1R34MH118314 (NIH)
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Mental Illness; Shared Decision Making
Keywords: serious mental illness; shared decision making-psychiatric medications; mental health
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coaching and Virtual Provider Group (Experimental): Mental Health Coaching and assigned practice with a Virtual Provider Program
  Interventions: Behavioral: Coaching and Virtual Provider Program Practice

INTERVENTIONS:
Behavioral: Coaching and Virtual Provider Program Practice — 4 weekly goal setting/coaching sessions, coupled with Virtual Provider program training and practice

SUMMARY:
GET PrEPD-Psychiatry is a mixed-methods, developmental study to adapt a shared decision making (SDM) intervention to be specific for psychiatry decisions (Aim 1, previously completed), evaluate its feasibility and acceptability (Aim 2), and examine potential mechanisms of change and preliminary outcomes (Aim 3) of this innovative intervention to increase SDM and self-management for adults with serious mental illness (SMI). In line with National Institute of Mental Health (NIMH) priorities, we are examining whether GET PrEPD-Psychiatry engages the target mechanisms that putatively underlie the intervention (i.e., patient activation and communication self-efficacy; Aim 3). Aim 1 used approximately 200 deidentified transcripts from our prior study of SDM in psychiatry to cull language used in decision-making. These conversations were then used to program the Virtual Provider to represent common interactions and decisions in psychiatric visits. Iterative testing of the use of the Virtual Provider has been completed and feedback was obtained from our psychiatry consultants to refine the program. For Aim 2, we will recruit up to 40 patients to participate in GET PrEPD-Psychiatry (4 weekly goal setting/coaching sessions, coupled with Virtual Provider training and practice). We will assess participant satisfaction and utility ratings, as well as track their use (frequency and time-on-task) of the Virtual Provider program. For Aim 3, we will follow enrolled patient participants, interviewing them at baseline and approximately 3 months later. We hypothesize that participants will have significantly 1) improved mechanisms of change, demonstrated by increases in self-reported activation and communication self-efficacy, 2) improved SDM, and 3) improved self-management and recovery attitudes. The Narrative Evaluation of Intervention Interview (NEII), completed at approximately 3 months, will be used as a qualitative interview guide to understand the acceptability and impact of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Current patient at the participating mental health center
* English speaking
* Willingness to participate in weekly coaching sessions, engage in practice with the Virtual Provider program

Exclusion Criteria:

* Under 18 years of age
* No reasonable access to use of internet on a computer
* Inability or unwillingness to use a computer (necessary for Virtual Provider Program practice)
* Never or rarely uses a computer or similar device (based on self-report)
* Very or somewhat uncomfortable using a computer or similar device (based on self-report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Salyers, PhD, Principal Investigator — Indiana University
Locations (1):
- Sandra Eskenazi Mental Health Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Coaching and Virtual Provider Group
Started | 29
Completed | 22
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Coaching and Virtual Provider Group
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
Primary Mental Health Diagnosis [Count of Participants; unit: Participants]
  Anxiety Disorders (Anxiety Disorder, Panic Disorder, Post-traumatic Stress Disorder) | 4
  Bipolar Disorder | 4
  Schizophrenia (Schizophrenia, Schizoaffective Disorder, Chronic Schizophrenia) | 12
  Major Depressive Disorder | 7
  Other (Difficulty Controlling Anger, Adjustment Disorder) | 2
Current Marital Status [Count of Participants; unit: Participants]
  Single, never married | 20
  Currently married or living with a partner | 2
  Separated or divorced | 6
  Widowed | 1
Highest Level of Education [Count of Participants; unit: Participants]
  Less than high school/GED | 5
  High school degree/GED | 9
  Some college coursework | 12
  Bachelors degree | 3
Current Employment Status [Count of Participants; unit: Participants]
  Paid Employment | 5
  Casual Work | 2
  Student | 1
  Unemployed and looking for work | 5
  Unemployed and not looking for work | 2
  Disabled | 13
  Other: Retired and Disabled | 1
Current Housing [Count of Participants; unit: Participants]
  Homeless (includes in shelter) | 3
  Staying with friends or family temporarily | 5
  Structured congregate living (e.g., nursing home, group home, residential facility) | 2
  Semi-independent living (staff member lives on site or foster family care) | 1
  Living with family (not spouse) | 4
  Own apartment or house-with spouse, living as married, with friends | 10
  Own apartment or house-alone | 4
Caretaking responsibilities for a child or children less than 18 years in same household [Count of Participants; unit: Participants]
  Yes | 5
  No | 24

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation Measure for Mental Health (PAM-MH)
Description: The 13-item Patient Activation Measure for Mental Health (PAM-MH) assesses patient knowledge, skill, and confidence for self-managing one's chronic health condition. Scores range from 0 to 100, with higher numbers indicating greater activation.
Time Frame: Baseline, 3 months
Population: 7 subjects were lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Virtual Provider Group
Number analyzed (Participants) | 29
units on a scale
  Baseline | 59.8 (17.1)
  3 Months: number analyzed (Participants) | 22
  3 Months | 61.6 (12.1)

2. Secondary Outcome: Altarum Consumer Engagement (ACE) Measure
Description: The 12-item Altarum Consumer Engagement (ACE) Measure assesses commitment, informed choice, and navigation. Scores range from 0-4, with higher scores indicating more engagement.
Time Frame: Baseline, 3 months
Population: 7 subjects were lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Virtual Provider Group
Number analyzed (Participants) | 29
units on a scale
  Baseline | 2.4 (0.7)
  3 Months: number analyzed (Participants) | 22
  3 Months | 2.4 (0.6)

3. Secondary Outcome: Perceived Efficacy in Patient-Provider Interactions (PEPPI-5)
Description: The 5-item Perceived Efficacy in Patient-Provider Interactions (PEPPI-5) measures patients' self-efficacy in obtaining medical information and getting their most important health concern discussed in a clinic visit; scores range from 1-10. The questionnaire is rated on a 10-point Likert scale, with higher scores indicating higher perceived efficacy in the interactions.
Time Frame: Baseline, 3 months
Population: 7 subjects were lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Virtual Provider Group
Number analyzed (Participants) | 29
units on a scale
  Baseline | 7.6 (2.1)
  3 Months: number analyzed (Participants) | 22
  3 Months | 7.4 (2.1)

4. Secondary Outcome: Illness Management and Recovery (IMR) Scale
Description: Illness self management will be assessed with the consumer-rated Illness Management and Recovery (IMR) Scale; items are rated on a 5-point behaviorally anchored scale and averaged. Scores range from 1 to 5, with higher number reflecting greater self-management.
Time Frame: Baseline, 3 months
Population: 7 subjects were lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Virtual Provider Group
Number analyzed (Participants) | 29
units on a scale
  Baseline | 3.4 (0.5)
  3 Months: number analyzed (Participants) | 22
  3 Months | 3.5 (0.5)

5. Secondary Outcome: Recovery Assessment Scale (Brief Version)
Description: Recovery attitudes will be assessed using the total score of the 20-item Brief version of the Recovery Assessment Scale. Using the average score, the scale ranges from 1 to 5, with 5 indicating greater self-reported recovery.
Time Frame: Baseline, 3 months
Population: 7 subjects were lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Coaching and Virtual Provider Group
Number analyzed (Participants) | 29
units on a scale
  Baseline | 4.0 (0.6)
  3 Months: number analyzed (Participants) | 22
  3 Months | 3.9 (0.5)

ADVERSE EVENTS:
Time Frame: approximately 3 months
Description: Adverse events were not systematically collected for this minimal risk study.
Arm/Group | Coaching and Virtual Provider Group
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04601194/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT04601194/ICF_001.pdf